CLINICAL TRIAL: NCT07326592
Title: A Phase 4, Multicenter, Double-blind, Study to Investigate the Efficacy, Safety, and Tolerability of 3 Active Doses of Respreeza® / Zemaira® Weekly Intravenous Infusions Administered Over 3 Years as Longterm Maintenance Therapy in Adult Subjects With Emphysema Related to Alpha1 Antitrypsin Deficiency
Brief Title: Phase 4, Double-blind Study Evaluating the Response on Computed Tomography (CT) Lung Density Decline Rates of Respreeza / Zemaira Weekly for 3 Years in Adults With alpha1 Antitrypsin Deficiency (AATD)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE1226_4003; 2025-522964-33-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-07; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-01

CONDITIONS: Alpha1 Antitrypsin Deficiency; Alpha1-Proteinase Inhibitor Deficiency; Emphysema
Keywords: Progressive Emphysema; Chronic Pulmonary Disease
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Emphysema | interventions — alpha 1-Antitrypsin; Respreeza

STUDY DESIGN:
Intervention Model Description: This is a double blind, parallel group assignment study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor will also be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CE1226 low dose (Active Comparator): CE1226 at low dose.
  Interventions: Biological: CE1226
- CE1226 medium dose (Experimental): CE1226 at medium dose.
  Interventions: Biological: CE1226
- CE1226 high dose (Experimental): CE1226 at high dose.
  Interventions: Biological: CE1226

INTERVENTIONS:
Biological: CE1226 — CE1226 will be administered via intravenous (IV) infusion weekly over 3 years.
  Other Names: Human alpha1-proteinase inhibitor; Respreeza; Zemaira

SUMMARY:
This is a multicenter, parallel-group, double-blind, randomized phase 4 study designed to identify the optimal dose of CE1226 (2 active doses) to slow disease progression as assessed by reduced rates of annual lung density decline in alpha-1 antitrypsin (AAT) deficient participants over 3 years as compared with the marketed dose 60 milligrams per kilogram (mg/kg).

ELIGIBILITY:
Inclusion Criteria:

* • Age greater than or equal to (>=) 18 and less than or equal to (<=) 65 years at the time of providing written informed consent.
* • Confirmed diagnosis of emphysema related to AATD with either the PiZZ, PiZ(null), or Pi(null/null) genotype with documented serum AAT levels less than (<) 11 micrometer (μM) (or < 50 mg/dL [milligram/deciliter]) at any time before the first administration of CE1226 on Day 1 (Baseline).

Exclusion Criteria:

* • Participants should not have acute illness or pulmonary exacerbation within 6 weeks before the first administration of CE1226 on Day 1 (Baseline).
* • Participants should not have previously received gene therapy for AATD at any point.
* • Participants with liver disease secondary to AATD.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2033-09-15 (Estimated); Study Completion 2033-09-15 (Estimated)

PRIMARY OUTCOMES:
Annual rate of change in adjusted lung density | From Baseline to Month 36
  The annual rate of change (expressed as gram per liter per year [g/L/year]) in adjusted lung density (15th percentile lung density [PD15]) will be calculated on CT scan assessments of whole lung at total lung capacity (TLC).

SECONDARY OUTCOMES:
Annual rate of change in forced expiratory volume in 1 second percent predicted (FEV1%) | From Baseline to Month 36
  The annual rate of change in FEV1% will be assessed by spirometry.
Annual rate of change in diffusion capacity of carbon monoxide (DLco) | From Baseline to Month 36
  The annual rate of change in DLco will be assessed by gas transfer using site machinery.
Number of severe pulmonary exacerbations | From screening up to Month 36
  Pulmonary excerbations will be assessed by the investigator using Rodriguez-Roisin criteria, where an exacerbation is defined as: a sustained worsening of the patient's condition, from a stable state and beyond normal day-to-day variations, necessitating a change in regular medication in a patient with underlying chronic obstructive pulmonary disease (COPD). A severe exacerbation is defined as an event requiring the introduction of corticosteroids and / or antibiotics which results in hospitalization or death.
Duration of severe pulmonary exacerbations | From screening up to Month 36
  Pulmonary excerbations will be assessed by the investigator using Rodriguez-Roisin criteria, where an exacerbation is defined as: a sustained worsening of the patient's condition, from a stable state and beyond normal day-to-day variations, necessitating a change in regular medication in a patient with underlying COPD. A severe exacerbation is defined as an event requiring the introduction of corticosteroids and / or antibiotics which results in hospitalization or death.
Number of participants experiencing treatment emergent adverse events (TEAEs) | From screening up to Month 36
Percentage of participants experiencing TEAEs | From screening up to Month 36

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (i.e. FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.